CLINICAL TRIAL: NCT05511610
Title: Accuracy of the MAAS Method (Minimal-flow Auto-control Anesthesia System) for the Administration of Desflurane and Sevoflurane in the Anesthetic Maintenance Phase. Prospective and Paired Observational Study.
Brief Title: MAAS Method (Minimal-flow Auto-control Anesthesia System) for the Administration of Desflurane and Sevoflurane
Acronym: MAAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAAS.Sevo.Desfl.accuracy
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Sevoflurane; Desflurane; Low Flow Anesthesia
Keywords: Sevoflurane; Desflurane; Anesthesia, Closed-Circuit
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAAS method trial (Experimental): Accuracy of sevoflurane and desflurane vaporizers to guarantee the ettHA%, based on the MAAS method.
  Interventions: Procedure: Sevoflurane uptake and supply; Procedure: Washout phase; Procedure: Desflurane uptake and supply; Procedure: Final phase

INTERVENTIONS:
Procedure: Sevoflurane uptake and supply — Phase sevo 1)
  * Moment 1 (M1): from OTI until end-tidal sevoflurane (etSEVO%) exceeds ettSEVO% by 10%. Deliver of sevoflurane to the system (SEVOdel) carried out by completely opening sevoflurane vaporizer (8%).
  * M2) once etSEVO% surpass ettSEVO% by 10%: turn off sevoflurane vaporizer and observe the progressive fall etSEVO%. When etSEVO% approaches ettSEVO% (0.1-0.2 points above ettSEVO%), the investigators will turn on the sevoflurane vaporizer following the MAAS method to ensure stability in inspired and expired concentrations of sevoflurane.
  Phase sevo 2) Objective: to maintain etSEVO% = ettSEVO% ±5% When the etSEVO% increases above the mentioned levels >> reduce SEVOdel by 0.25-0.5%.
  When the etSEVO% decreases below the mentioned levels>> increase SEVOdel by 0.25-0.5%.
Procedure: Washout phase — The investigators will close the sevoflurane vaporizer and will start the administration of Propofol in intravenous perfusion; the investigators will then open the FGF sequentially at 2>5>10 liters per minute (LPM), until the etSEVO% is <0.2 MAC.
Procedure: Desflurane uptake and supply — Phase desflu 1)
  * Moment 1 (M1): from the end of Washout phase until end-tidal desflurane (etDESFLU%) exceeds ettDESFLU% by 10%. Deliver of desflurane to the system (DESFLUdel) carried out by completely opening the desflurane vaporizer (18%).
  * M2) once etDESFLU% surpass ettDESFLU% by 20%: turn off the desflurane vaporizer and observe the progressive fall etDESFLU%. When etDESFLU% approaches ettDESFLU% (0.8-1.2 points above ettDESFLU%), the investigators will turn on the desflurane vaporizer following the MAAS method to ensure stability in inspired and expired concentrations of desflurane.
  Phase desflu 2) Objective: to maintain etDESFLU% = ettDESFLU% ±5% When the etDESFLU% increases above the mentioned levels >> reduce DESFLUdel by 0.25-0.5%.
  When the etDESFLU% decreases below the mentioned levels>> increase DESFLUdel by 0.25-0.5%.
Procedure: Final phase — From the end of Phase desflu 2 until the end of the intervention. Maintenance of anesthesia with desflurane following the principles of MAAS Method.
  Between 15-20 minutes before the end of the intervention, the investigators will stop the administration of desflurane, registering the time until the reaching etDESFLU% < 0.2 MAC.

SUMMARY:
In the present work the investigators will study the accuracy of the MAAS (Minimal-flow Autocontrol Anesthesia System) method to estimate the percentage of halogenated anesthetic (HA) to be supplied to the anesthetic circuit based on the estimation of HA uptake during the maintenance phase. The investigators will evaluate the accuracy of sevoflurane and desflurane vaporizers to guarantee the administration of that amount of estimated HA, thus guaranteeing the maintenance of the target concentration of HA at the end of expiration: end-tidal target HA% (ettHA%). To do this, the investigators will quantify the number of adjustments that need to be made to each vaporizer to maintain ettHA%. As secondary objectives, the investigators will analyze the time to reach the target concentration of HA, the deviations that occur from that concentration despite the correct application of the method, and the consumption of HA during the procedure.

Through the entire procedure, all participants will be ventilated under a tailored open lung approach (tOLA) strategy.

DETAILED DESCRIPTION:
Halogenated anesthetics (HAs) are the gaseous drugs commonly used in inhalation anesthesia to ensure, among other effects, loss of consciousness or induction of "anesthetic sleep". They are administered in their gaseous state through the anesthesia vaporizers inserted in the anesthesia workstations. Like other gaseous hydrocarbons, HAs contribute to global warming, with the particularity that their global warming potential (GWP) is hundreds of times higher than that of the reference molecule, CO2, especially in the case of desflurane. For this reason, professionals and administrations must be especially sensitive when handling this type of drugs. Indeed, the investigators consider that its use should be questioned in the absence of administration devices capable of minimizing atmospheric emissions, provided that there are adequate therapeutic alternatives.

Currently, there are "universally" available tools that guarantee that these minimum contamination principles can be met in daily practice. The fundamental tool would be the anesthesia circle breathing circuit. Circle circuits are conceived as artificial breathing systems that allow the rebreathing of exhaled gases. Rebreathing exhaled gases, once the CO2 has been removed by means of gas neutralization systems incorporated in anesthesia stations (CO2 absorbers), is safe and effective, and today this mode of administration of the inhalation anesthesia has become the gold standard. The usefulness and efficiency of circle circuits is anesthesiologist-dependent, since the reuse of exhaled gases will depend on the amount of "new" (fresh) medicinal gases that the anesthesiologist allows to enter the anesthesia workstation every minute, by means of the regulation of the fresh gas flow (FGF): the higher FGF, the less reuse of exhaled gases and at the greater surplus of "waste" gases to be evacuated and expelled into the atmosphere. On the contrary, the fewer new gases the anesthesiologist allows to enter the anesthesia workstation, the greater the reuse of exhaled gases, and the smaller the volume of gases expelled into the atmosphere. The administration of inhalation anesthesia through the use of low FGF, known as low flow anesthesia (LFA) techniques, would therefore constitute one of the main contributors to the reduction of HA emissions into the atmosphere.

The majority of anesthesia workstations used in daily practice allow anesthesiologists to work with FGF lower than 500 milliliters per minute (ml/min) or reaching to the closed-circuit anesthesia mode, that modality of inhalation anesthesia in which it is supplied to the system (anesthesia workstation and patient) the amount of gases (ml/min) that are transferred ("lost") from the central compartment (blood and highly perfused organs- HPO) to other compartments due to the principle of partial pressures equilibrium between different compartments (uptake phenomenon by muscle and fat), or metabolic consumption in the case of O2.

Different techniques for administering LFA have been described. The MAAS method (Minimal-flow Autocontrol Anesthesia System) proposes a didactic and easy way to estimate the needs for HA supplementation during the anesthetic maintenance phase, and includes a feasible formulation when adjusting the supply of HA to the system. The maintenance phase would comprise from the moment in which the target concentration of HA in the central compartment is reached, until the moment in which HA stops being administered to the system. During this period, HA keeps on being transferred towards muscle and fat from the central compartment (highly perfused organs (HPO) compartment) following the principle of partial pressures equilibrium. The estimation of HA uptake (HAup) by muscle and fat once the equilibrium state between the anesthesia workstation (respiratory circuit) and the HPO is reached, is based on the calculation HAup (ml/min) =HAfi-HAfe*MV(ml/min), where HAfi and HAfe state for inspired and expired fraction of HA, respectively; and MV for volume minute.

The estimate of the ml of HA to be supplied to the anesthetic circuit through the FGF, would be done following the formula HAdel (from HA delivered)= HAup (ml/min )*100% /FGF(ml).

The main objective of this work will be to compare the accuracy of sevoflurane and desflurane vaporizers to guarantee the ettHA% based on the MAAS method, which will be quantified based on the number of adjustments that must be made in each vaporizer to maintain the predefined ettHA% As secondary objectives, the investigators will analyze the time to reach the ettHA%, the deviations that occur from that ettHA% despite the correct application of the method, and the consumption of HA (ml of HA in its liquid phase) during the procedure

METHODS Prospective, paired, observational study with consecutive recruitment of participants to be carried out in a tertiary care teaching hospital (Hospital Universitario Virgen del Rocío, Sevilla). Approval for this study will be sought from the local ethics committee (Ethics Committee of the Hospital Universitario Virgen del Rocío y Virgen Macarena, Seville), and the study will be registered in Clinical Trials prior to the start of recruitment (http://www.clinicaltrials .gov.) Study design Those adult subjects (≥ 18 years) scheduled for robotic urological, coloproctological or gynecological surgery in the investigators´ institution will be included after obtaining the corresponding written informed consent. The participants will be recruited consecutively depending on the availability of the researchers until the estimated sample is completed. Exclusion criteria are detailed in the "Eligibility" section of this document.

Study protocol On the day of surgery, standard monitoring will begin upon arrival in the operating room, including electrocardiography, pulse oximetry, and non-invasive blood pressure monitoring. After conscious sedation with intravenous (IV) midazolam 1 to 2 mg and remifentanil infused 0.03-0.05 µg/kg/min, participants will be pre-oxygenated through a face mask for 5 min under spontaneous ventilation with an inspired fraction of oxygen (FIO2) of 0.8 and a FGF of 6 L/min. General anesthesia will be induced with propofol (1-1.5 mg/kg of predicted body weight [PBW]), administer 0.8 mg/kg rocuronium PBW, and proceed with orotracheal intubation (OTI). Patients will be ventilated through a Primus anesthesia workstation (Drager, Telford, PA, USA) using a tidal volume (TV) of 7 mg*kg-1 PBW. The ventilatory mode used will be volume control, using a tailored open lung approach (tOLA) protective pulmonary ventilation strategy (see below) that will include an inspiration:expiration ratio of 1:2 and a respiratory rate of 12-15 breaths/min to maintain an end-tidal CO2 (etCO2) between 35 and 40 mmHg and an initial PEEP of 5 cmH2O (10 cmH2O in the case of BMI > 30). A 30% inspiratory pause will be scheduled for all participants. A FGF corresponding with the 10% of minute volume with an inspired FIO2 of 0.5 will be used throughout the procedure. Anesthesia will be maintained with remifentanil 0.03 to 0.05 µg/kg/min and sevoflurane or desflurane, depending on the phase of the study.

Initially sevoflurane will be used, with a minimum alveolar concentration (MAC) ranging from 0.7 to 0.8 adjusted to the patient's age (predefined MAC), to guarantee a Bispectral Index (BIS Quatro; Covidien Ilc, Mansfield, MA, USA) between 40-60. The investigators will establish as an objective for anesthetic maintenance an ettHA% that will correspond to the predefined MAC and will be the parameter used as a reference throughout the study. Rocuronium will be administered to ensure deep neuromuscular blockade during the procedure, and will be monitored by train of four neuromuscular relaxation (TOF-watch®, Organon Ltd., Swords, Co. Dublin, Ireland). Other drugs that will be systematically used enclose dexamethasone 8 mg IV after induction, paracetamol 1 g after induction and 1 g at the end of the procedure (in surgeries lasting > 2 h); dexketoprofen 50 mg at the end of surgery. Ondansetron 8 mg prior to eduction; and local anesthesia with 0.25% bupivacaine on the access ports. All ventilation parameters will remain stable throughout the study except PEEP, which will be adapted according to tOLA ventilation principles.

Tailored Open Lung Approach strategy The base of this strategy will be: 1) TV of 7 ml/kg of ideal weight (PBW, of the English predicted body weight); 2) performing a systematic alveolar recruitment maneuver (ARM) following the model of Tusman and Ferrando; 3) the use of individualized and optimized positive end expiratory pressure (PEEP), understood as that which guarantees greater compliance of the respiratory system after ARM.

Statistical analysis Statistical analysis will be performed by the principal investigator. For data analysis, the statistical software IBM SPSS Statistics for Windows, version 24 (IBM Corp., Armonk, NY, USA) will be used. The investigators will perform an exploratory analysis of the data, using the mean ± standard deviation or the median with interquartile range for quantitative variables, and will use percentages for the analysis of qualitative variables. The investigators will check the normality of data distribution with the Kolmogorov-Smirnov test or with the Shapiro-Wilk test for variables with less than 50 records. The Student's t test for paired samples will be used to study the behavior of the quantitative variables at different times (intragroup comparisons). To compare intragroup qualitative variables, the Wilcoxon test for paired samples will be used.

Sample's size calculation To calculate the size of the sample, version 4.2 of the statistical program EPIDAT (General Directorate of Innovation and Public Health Management of the Ministry of Health of the Junta de Galicia) will be used. The minimum required sample will be determined based on the results of the study on a pilot sample of 5 paired cases (1st sevoflurane and 2nd desflurane) in which the number of precise changes in the vaporizer to guarantee the stability of the ettHA% will be determined. The sample size will be calculated to obtain a power of 80% to detect differences in the contrast of the null hypothesis h₀: μ₁ = μ₂ using a two-sided Student's t-test for two related samples, considering a level of significance of 5% and assuming the respective standard deviation in each group.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 18 years) scheduled for robotic urological, coloproctological or gynecological surgery in the investigators´ institution
* Written informed consent

Exclusion Criteria:

* Participation in another interventional study
* Participants unable to understand the information contained in the informed consent
* American Society of Anesthesiologists (ASA) classification grade = IV
* Patient in dialysis
* Chronic obstructive pulmonary disease (COPD) grade Global Initiative for Chronic Obstructive Lung Disease(GOLD) > 2
* Functional vital capacity < 60% or > 120% of the predicted
* Body mass index (BMI) > 35 kg/m2
* New York Heart Association (NYHA) functional class ≥ 3
* Clinically suspected heart failure
* Diagnosis or suspicion of intracranial hypertension
* Presence of pneumothorax or giant bullae on preoperative imaging tests
* Use of Continuous Positive Airway Pressure (CPAP).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Changes made in the sevoflurane vaporizer | 60 minutes, starting from the end of Phase sevo 1 (once filled the HPO compartment)
  Number of adjustments that must be made in the sevoflurane vaporizer to maintain the predefined end-tidal target of sevoflurane (ettSEVO%).
Changes made in the desflurane vaporizer | 60 minutes, starting from the end of Phase desflu 1(once filled the HPO compartment)
  Number of adjustments that must be made in the desflurane vaporizer to maintain the predefined end-tidal target of desflurane (ettDESFLU%).

SECONDARY OUTCOMES:
Time to reach the ettSEVO% | Immediately after OTI and until completing the Phase sevo 1
  Time (minutes) to reach the ettSEVO%; measured from the time of OTI until completing the Phase sevo 1. Includes M1 and M2 of this Phase.
Time to reach the ettDESFLU% | Immediately after completing the Washout phase and until completing the Phase desflu 1.
  Time (minutes) to reach the ettDESFLU%; measured from the starting of Phase desflu 1 until completing this Phase desflu 1. Includes M1 and M2 of this Phase.
Deviations from ettSEVO% despite the correct application of the method | 60 minutes: starting from the end of Phase sevo 1 until the end of Phase sevo 2
  Deviations that occur from that ettSEVO% despite the correct application of the method.
  Following the modified Wetz model, all the time periods in which the HA is outside the target range will be recorded, as well as the percentage of deviation over that range. Then, the investigators will calculate the duration of those periods with deviated values with respect to the total duration of the measured phase. The accuracy and stability of the method will be established based on the duration of these periods and their magnitude (degree of deviation) with respect to the study phase.
Deviations from ettDESFLU% despite the correct application of the method | 60 minutes: starting from the end of Phase desflu1 until the end of Phase desflu 2
  Following the modified Wetz model, all the time periods in which the HA is outside the target range will be recorded, as well as the percentage of deviation over that range. Then, we will calculate the duration of those periods with deviated values with respect to the total duration of the measured phase. The accuracy and stability of the method will be established based on the duration of these periods and their magnitude (degree of deviation) with respect to the study phase.
Consumption of HA (ml of HA in its liquid phase) during the procedure | During the procedure: starting pre-intervention and immediately after the procedure
  To estimate the consumption of ml of liquid HA, the investigators will calculate the difference in weight of the vaporizer before and after procedure in each case, using a precision scale and taking into account the density and specific weight specifications set by the manufacturer for sevoflurane and desflurane.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel de la Matta, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

REFERENCES:
- [Background] McGain F, Muret J, Lawson C, Sherman JD. Environmental sustainability in anaesthesia and critical care. Br J Anaesth. 2020 Nov;125(5):680-692. doi: 10.1016/j.bja.2020.06.055. Epub 2020 Aug 12. PMID 32798068
- [Background] Sherman J, Le C, Lamers V, Eckelman M. Life cycle greenhouse gas emissions of anesthetic drugs. Anesth Analg. 2012 May;114(5):1086-90. doi: 10.1213/ANE.0b013e31824f6940. Epub 2012 Apr 4. PMID 22492186
- [Background] Petre MA, Malherbe S. Environmentally sustainable perioperative medicine: simple strategies for anesthetic practice. Can J Anaesth. 2020 Aug;67(8):1044-1063. doi: 10.1007/s12630-020-01726-0. Epub 2020 Jun 8. PMID 32514694
- [Background] Brattwall M, Warren-Stomberg M, Hesselvik F, Jakobsson J. Brief review: theory and practice of minimal fresh gas flow anesthesia. Can J Anaesth. 2012 Aug;59(8):785-97. doi: 10.1007/s12630-012-9736-2. Epub 2012 Jun 1. PMID 22653840
- [Background] Carter LA, Oyewole M, Bates E, Sherratt K. Promoting low-flow anaesthesia and volatile anaesthetic agent choice. BMJ Open Qual. 2019 Sep 13;8(3):e000479. doi: 10.1136/bmjoq-2018-000479. eCollection 2019. PMID 31637316
- [Background] Colak YZ, Toprak HI. Feasibility, safety, and economic consequences of using low flow anesthesia according to body weight. J Anesth. 2020 Aug;34(4):537-542. doi: 10.1007/s00540-020-02782-y. Epub 2020 May 3. PMID 32363423
- [Background] Ferrando C, Suarez-Sipmann F, Tusman G, Leon I, Romero E, Gracia E, Mugarra A, Arocas B, Pozo N, Soro M, Belda FJ. Open lung approach versus standard protective strategies: Effects on driving pressure and ventilatory efficiency during anesthesia - A pilot, randomized controlled trial. PLoS One. 2017 May 11;12(5):e0177399. doi: 10.1371/journal.pone.0177399. eCollection 2017. PMID 28493943
- [Background] Tusman G, Groisman I, Fiolo FE, Scandurra A, Arca JM, Krumrick G, Bohm SH, Sipmann FS. Noninvasive monitoring of lung recruitment maneuvers in morbidly obese patients: the role of pulse oximetry and volumetric capnography. Anesth Analg. 2014 Jan;118(1):137-44. doi: 10.1213/01.ane.0000438350.29240.08. PMID 24356163
- [Background] Wetz AJ, Mueller MM, Walliser K, Foest C, Wand S, Brandes IF, Waeschle RM, Bauer M. End-tidal control vs. manually controlled minimal-flow anesthesia: a prospective comparative trial. Acta Anaesthesiol Scand. 2017 Nov;61(10):1262-1269. doi: 10.1111/aas.12961. Epub 2017 Aug 22. PMID 28832896